RESEARCH PROTOCOL - Use of the eFisioTrack system for monitoring prescribed therapeutic exercises in patients with shoulder orthopedic injuries in a hospital setting: A pilot feasibility study

5 6

# PROJECT SUMMARY

7 8

9

#### Rationale

To assess the effects of the eFisioTrack monitoring system on clinical variables in patients with prescribed physiotherapy for shoulder injuries.

10 11 12

# **Objectives**

The main aim of the study was to evaluate the effect on clinical variables of monitoring exercises prescribed for shoulder injury rehabilitation with the eFisioTrack platform in patients of the Rehabilitation Service at University Hospital of Elche.

1617

# Methods

- A pilot feasibility study, single bling with two groups (experimental and control group).
- 19 Clinical outcome measures will be shoulder function and pain (Constant Murley Score
- and Disabilities of the Arm, Shoulder, and Hand or DASH score). Each variable will be
- 21 measured by a blinded physiotherapist at baseline and at one month follow-up. Patients
- 22 performed the prescribed exercises either supervised by the physiotherapist (control
- group) or in a separate room without therapist supervision (experimental group).

2425

# **Population**

The study will be carried out in the buildings of the Rehabilitation Service at University Hospital of Elche, starting in July 2023 and finishing in December 2023.

28

# 29 Expected outcomes.

- 30 This study aims to contribute to the advancement of the knowledge about the shoulder
- 31 treatment. The system shows promising results as a work item in shoulder home-based
- 32 rehabilitation. In fact, real-time telerehabilitation is a strategy for interventions in other
- 33 musculoskeletal conditions, to provide continuity to healthcare services and mitigate
- 34 distance and displacements. Confirmation of these preliminary results could reduce the
- workload of physiotherapy services, contributing to resource efficiency.

3637

#### GENERAL INFORMATION

- 38 Protocol title. Use of the eFisioTrack system for monitoring prescribed therapeutic
- 39 exercises in patients with shoulder orthopedic injuries in a hospital setting: A pilot
- 40 feasibility study.
- 41 **Protocol identifying number.** The study protocol was approved by the Ethics and
- 42 Research Committee of General University Hospital of Elche (CEIC HGUE-Shs2011).
- 43 **Registration date.** 21/07/2014
- Name and address of the sponsor/funder. This research received no external funding.

# 1 Investigator responsible

# 2 Research site.

# 3 Authors.

6

9

4 (Ensure the names of research participants are not included in an uploaded document).

#### **Author Contributions:**

7 (Ensure the names of research participants are not included in an uploaded document).

# RATIONALE AND BACKGROUND INFORMATION

- 10 Shoulder pain is a common health problem, and its prevalence has been estimated at
- around 7%–26%. There are several conditions that can produce pain in the shoulder
- 12 complex, such as fractures, frozen shoulder, rotator cuff tendinopathy, or subacromial
- syndrome. Physiotherapy management helps to reduce pain, improve range of movement
- and strength, and improve function. Combining active exercises with manual therapies is
- a common practice when treating musculoskeletal injuries of the shoulder.
- 16 Therapeutic exercise, in both the physical therapy setting and at home, is a fundamental
- 17 component of shoulder rehabilitation plans whether treatment is performed with or
- without surgery, and there is evidence of its effectiveness in the management of shoulder
- 19 conditions<sup>5</sup>. The primary goal of a shoulder exercise program is to relieve pain, increase
- 20 strength, reduce muscle imbalances, and restore pain-free joint range of motion.
- 21 Therefore, its correct execution is of great importance for the clinical course.
- 22 However, one of the main problems in orthopedic shoulder rehabilitation is poor
- 23 adherence to home exercise prescriptions. Some strategies for their control, such as daily
- or video recording, have been described, but their use is limited by recall bias or the need
- 25 for advanced technology.
- 26 There is a growing number of trials about the use of technology to monitor rehabilitation
- exercises. Its application in shoulder injuries could be potentially beneficial. Carbonaro
- 28 et al. presented the development and preliminary testing of a wearable-technology
- 29 platform for the remote rehabilitation of shoulder muscular-skeletal diseases. This system
- 30 (Shoulphy) was designed to lead and assess the patient wearing a minimal set of inertial
- 31 sensors and following personalized physical rehabilitation programs under the remote
- 32 supervision of the physician/therapist. Pan et al. reported the use of accelerometer-based
- 33 sensors built into a smartphone to capture the rehabilitation exercises as a self-home
- monitoring system. Wearable sensors, smartphones, and inertial measurement units have
- become a feasible option for monitoring joint movement. There is also research on the
- 36 application of Nintendo® Wii-technology for monitoring therapeutic exercises on
- 37 shoulder injuries<sup>16</sup>. This is based on accelerometers and gyroscopes located in the
- 38 controls, making it a low-cost option. However, most of these focus on stroke, to improve
- 39 arm function and balance in hemiparetic patients
- 40 Ruiz-Fernandez et al. described a software platform based on Wii-controls technology
- 41 that could be used to monitor patients' activity in the scheduled exercise sessions.
- However, there is no clinical study of the results obtained in the laboratory. Therefore,
- 43 the aim of this pilot study was to evaluate the effect on clinical variables of monitoring
- 44 exercises prescribed for shoulder injury rehabilitation with the eFisioTrack platform in
- 45 patients of the Rehabilitation Service at University Hospital of Elche.

#### **OBJECTIVES**

- The main aim of the study was to evaluate the effect on clinical variables of monitoring exercises prescribed for shoulder injury rehabilitation with the eFisioTrack platform in
- 5 patients of the Rehabilitation Service at University Hospital of Elche.

6

7

STUDY DESIGN

- 8 A pilot feasibility study, single bling with two groups (experimental and control group).
- 9 Clinical outcome measures will be shoulder function and pain (Constant Murley Score
- and Disabilities of the Arm, Shoulder, and Hand or DASH score). Each variable will be
- measured by a blinded physiotherapist at baseline and at one month follow-up. Patients
- 12 performed the prescribed exercises either supervised by the physiotherapist (control
- group) or in a separate room without therapist supervision (experimental group).

14 15

# Regarding the study population.

- Patients who will be referred to the rehabilitation service of the University Hospital of
- 17 Elche (Spain) for physiotherapy treatment (manual therapy, exercise, stretching, and
- electrotherapy) after suffering orthopedic injury or surgery in the shoulder joint complex,
- 19 from July 2023 to December 2023 will be considered for enrollment in the study.

# 20 Inclusion criteria were established as follows:

- (i) be at least 18 years old and be able to read and understand Spanish.
- (ii) suffer a traumatic or degenerative shoulder injury, with or without surgical treatment.
- (iii) have a prescription for rehabilitative physical therapy that includes active exercises.

25 26

21

22

23

24

2627

28

# The exclusion criteria adopted were:

Patients were excluded if they had a concomitant injury on an upper extremity or the cervical spine at the time of participation or sequelae of previous injuries in the area.

293031

# Regarding sample size

- The main objective of this study is to know whether a clinical trial will be feasible and to
- have an estimate of standard deviation, which will be used in the sample size calculation
- for the large-scale trial; to estimate the rate (proportion) of eligible people who are willing
- to participate, of participants who drop out of the trial, or of participants who comply with
- 36 the assigned intervention. That is why the sample size could be between 20 and 40
- 37 participants.

38

39

# METHODOLOGY

- 40 Following baseline examination, patients will be randomly assigned to either
- 41 physiotherapist-supervised exercise (control group) or monitoring by the eFisioTrack

- 1 system (experimental group). Patients will perform the prescribed exercises either
- 2 supervised by the physiotherapist (control group) or in a separate room without therapist
- 3 supervision (experimental group). A system of codes (four last numbers of the patient's
- 4 ID number) was assigned to each participant using a computerized application (Research
- 5 randomizer: www.randomizer.org). Clinical outcome measures were shoulder function
- 6 and pain (Constant Murley Score and Disabilities of the Arm, Shoulder, and Hand or
- 7 DASH score). Each variable was measured by a blinded physiotherapist at baseline and
- 8 at one month follow-up.
- 9 The intervention consists of the use of the eFisioTrack platform in the experimental group
- 10 to perform active exercises as part of their shoulder rehabilitation. These were performed
- independently by each patient in a hospital room, using the efisioTrack system without
- supervision by the physiotherapist. The design and use of eFisioTrack has been assessed
- for usability and was described as appropriate and technically feasible. The subjects will
- be previously instructed in the use of the system in two 20-minute sessions. The type of
- exercise and its parameters will be chosen and progressed considering the functional
- status of the patient and being similar to those executed under the physiotherapist's
- 17 supervision.

# **OUTCOME MEASURES**

- 20 The baseline measures will be collected before randomization and the outcome
- 21 assessments will blind. All assessment measures, will be collected by the same clinician
- 22 who was not involved in the treatment programs. In addition, at the physiotherapy service
- patients received a paper copy of the questionnaires to fill out on their own.
- 24 The following patient-reported outcome measures were used to assess participants'
- 25 shoulder pain and function: the Disabilities of Arm, Shoulder and Hand (DASH) score
- and the Constant-Murley (CM) score.

# 27 • Primary outcome measures

- 28 The DASH was taken as a primary outcome measure. It is one of the most widely used
- 29 self-reported questionnaires that measures symptoms and degree of function related to a
- disorder in the upper extremity. It has been validated in Spanish and comprises 30 items:
- 31 21 about physical function, 6 for symptoms, and 3 to assess social aspects. In addition,
- there are two optional modules, each with four items, which are used to assess symptoms
- and function in those whose functional demands are not included in the main part of the
- 34 questionnaire.
- 35 This instrument has been used in previous studies involving physical therapy and exercise
- 36 for shoulder injuries. It is scored in two components: first the symptom questions (30
- items) and second the optional modules. The assigned values for all completed responses
- are summed and averaged, producing a score that is then transformed on a scale of 0 to
- 39 100 by subtracting one and multiplying by . A higher score indicates greater disability.
- 40 Differences in scores are considered clinically relevant (minimum clinically important
- 41 difference or MCID) when they are above 10 points.

# 42 • Secondary outcome measures

- The CM score is a commonly used specific instrument for assessing the shoulder joint.
- The maximum score is 100 points, 90 to 100 being excellent, 80 to 89 good, 70 to 79

- 1 medium, and less than 70 poor, considering that the scores can vary with age. This tool
- 2 includes a subjective assessment of the patient's pain and ability to perform daily
- 3 activities (35 points) and an objective assessment of mobility and strength by physical
- 4 examination (65 points). Its use has been specifically validated in shoulder arthroplasty,
- 5 rotator cuff repair, adhesive capsulitis, and fractures of the proximal humerus, but not in
- 6 shoulder instability.

# SECURITY CONSIDERATION

- 9 The risks of the treatment techniques or manual therapy procedures as well as other means
- of physical treatment and their possible adverse effects that will be used in this study are
- 11 uncommon and generally mild. Follow-up of cases with adverse effects will be
- maintained until the end of the study. This measure ensures safe conditions for the
- 13 treatment of patients.

1415

# STATISTICAL ANALYSIS

- 16 Descriptive data will be presented as a mean and standard deviation for continuous
- variables. For statistical analyses, the normality of the data distribution will be assessed
- by the Shapiro-Wilk test. To compare differences between groups in the studied variables,
- 19 the Student's t-test will be used for normally distributed data. For each group, a paired t-
- 20 test will be used to compare baseline and follow-up scores, and the 95% confidence
- 21 interval (CI) will be calculated for the mean differences.
- 22 The theoretical sample size based on a 10-point difference (10%) in the DASH between
- 23 the two studied groups, assuming a 95% confidence interval, 80% statistical power and
- 24 20% sampling error, resulted in 36 patients in each group.
- 25 All analyses will be conducted using SPSS Statistical Package for Windows, version 25
- 26 (SPSS Inc., 2009, Chicago, Illinois, USA). The significance level was set at P < 0.05.

27

28

# EXPECTED OUTCOMES OF THE STUDY

- 29 This study aims to contribute to the advancement of the knowledge about the treatment
- 30 of acute grade II WL, showing the effectiveness of SAT technique compared to other
- 31 frequently used treatment protocols. The lack of randomized clinical trials related to the
- 32 application of spinal manipulation techniques in whiplash injury, compared to studies in
- which passive and active interventions are applied, increases the interest of this study.

3435

# PROJECT DURATION

- 36 The study will be carried out in the buildings of the Rehabilitation Service at University
- Hospital of Elche, starting in July 2023 and finishing in December 2023.

38

39

# ETHICAL ASPECTS

- 1 The study protocol was approved by the Ethics and Research Committee of General
- 2 University Hospital of Elche (CEIC HGUE-Shs2011). All participants will sign an
- 3 informed consent form prior to voluntary participation in the study.
- 4 The ethical requirements relevant to patient safety, as set out in the Declaration of
- 5 Helsinki and the Belmont Report on Respect for Persons will be followed during the
- 6 study. Furthermore, the patient will sign the informed consent form to authorise his or her
- 7 inclusion in the study, confirming beforehand that he or she understood the study
- 8 correctly.

# REFERENCES

11

- 12 1. Lucas J, van Doorn P, Hegedus E, Lewis J, van der Windt D. A systematic review of the global prevalence and incidence of shoulder pain. BMC Musculoskelet
- Disor. 2022;23(1):1073. doi: 10.1186/s12891-022-05973-8.
- 2. Greenberg DL. Evaluation and treatment of shoulder pain. Med Clin North Am. 2014
- 16 May;98(3):487-504. doi: 10.1016/j.mcna.2014.01.016.
- 3. Paje MJ, Green S, McBain B, Surace SJ, Deitch J, Lyttle N, Mrocki MA, Buchbinder
- R. Manual therapy and exercise for rotator cuff disease. Cochrane Database Syst
- 19 Rev. 2016;2016(6):CD012224. doi: 10.1002/14651858.CD012224.
- 4. Kromer TO, Tautenhahn UG, de Bie RA, Staal JB, Bastiaenen CH. Effects of
- 21 physiotherapy in patients with shoulder impingement syndrome: a systematic review
- of the literature. J Rehabil Med. 2009;41(11):870-80. doi: 10.2340/16501977-0453.
- 5. Babatunde O, Ensor J, Littlewood C, Chesterton L, Jordan JL, Corp N, Wynne-
- Jones G, Roddy E, Foster NE, van der Windt DA. Comparative effectiveness of
- 25 treatment options for subacromial shoulder conditions: a systematic review and
- 26 network meta-analysis. Ther Adv Musculoskelet
- 27 Dis. 2021;13:1759720X211037530. doi: 10.1177/1759720X211037530.
- 28 6. Paraskevopoulos E, Plakoutsis G, Chronopoulos E, Maria P. Effectiveness of
- 29 Combined Program of Manual Therapy and Exercise Vs Exercise Only in Patients
- With Rotator Cuff-related Shoulder Pain: A Systematic Review and Meta-analysis.
- 31 Sports Health. 2022;19417381221136104. doi: 10.1177/19417381221136104.
- 7. Holgrem T, Hallgren HB, Öberg B, Adolfsson L, Johansson K. Effect of specific
- 33 exercise strategy on need for surgery in patients with subacromial impingement
- 34 syndrome: randomised controlled study. BMJ. 2012; 20;344:e787. doi:
- 35 10.1136/bmj.e787.
- 8. Burns D, Boyer P, Razmjou H, Richards R, Whyne C. Adherence Patterns and Dose
- Response of Physiotherapy for Rotator Cuff Pathology: Longitudinal Cohort Study.
- 38 JMIR Rehabil Assist Technol. 2021;8(1):e21374. doi: 10.2196/21374.
- 9. Bassett SF. The assessment of patient adherence to physiotherapy rehabilitation. NZ
- 40 J Physiother 2003; 31(2): 1-6.

- 1 10. Baroni MP, Jacob M, Rios WR, Fandim JV, Fernandez LG, Chaves PI, Fioratti I,
- 2 Saragiotto BT. The state of the art in telerehabilitation for musculoskeletal
- 3 conditions. Arch Physiother. 2023;13(1):1. doi: 10.1186/s40945-022-00155-0.
- 4 11. Eriksson L, Lindström B, Ekenberg L. Patients' experiences of telerehabilitation at
- 5 home after shoulder joint replacement. J Telemed Telecare 2011; 17(1): 25-30. doi:
- 6 10.1258/jtt.2010.100317
- 7 12. Carbonaro N, Lucchesi I, Lorusssi F, Tognetti A. Tele-monitoring and tele-
- 8 rehabilitation of the shoulder muscular-skeletal diseases through wearable systems.
- 9 Annu Int Conf IEEE Eng Med Biol Soc. 2018:4410-4413. doi:
- 10 10.1109/EMBC.2018.8513371.
- 13. Pan JI, Chung HW, Huang JJ. Intelligent Frozen Shoulder Self-Home Rehabilitation
- Monitoring System. Proceedings, The 2nd International Conference on Information
- 13 Science and Technology. IST 2013, ASTL Vol. 23, pp. 265 270, 2013.
- 14. Carnevale A, Longo UG, Schena E, Massaroni C, Lo Presti D, Berton A, Candela V,
- Denaro V. Wearable systems for shoulder kinematics assessment: a systematic
- review. BMC Musculoskelet Disord. 2019;20(1):546.doi: 10.1186/s12891-019-
- 17 2930-4. PMID: 31731893; PMCID: PMC6858749.
- 18 15. Sliepen M, Lipperts M, Tjur M, Mechlenburg I. Use of accelerometer-based activity
- monitoring in orthopaedics: benefits, impact and practical considerations. EFORT
- 20 Open Rev. 2020;4(12):678-685. doi: 10.1302/2058-5241.4.180041.
- 21 16. Rizzo JR, Thai P, Li E, Tung T, Hudson TE, Herrera J, Raghavan P. Structured Wii
- 22 protocol for rehabilitation of shoulder impingement syndrome: A pilot study. Ann
- 23 Phys Rehabil Med 2017;60(6):363-370. doi: 10.1016/j.rehab.2016.10.004.
- 24 17. Anwar N, Karimi H, Ahmad A, Gilani S, Khalid K, Aslam A, Hanif A. Virtual
- 25 Reality Training Using Nintendo Wii Games for Patients With Stroke: Randomized
- 26 Controlled Trial. JMIR Serious Games. 2022; 10(2):e29830. doi: 10.2196/29830.
- 27 18. Adie K, Schofield Ch, Berrow M, Wingham J, Humfryes J, Pritchard C, James M,
- Allison R. Does the use of Nintendo Wii Sports<sup>TM</sup> improve arm function? Trial of
- Wii<sup>TM</sup> in Stroke: a randomized controlled trial and economics analysis.Clin Rehabil.
- 30 2017; 31(2):173-185. doi: 10.1177/0269215516637893.
- 31 19. Ruiz-Fernández D, Marín-Alonso O, Soriano-Paya A, García-Pérez JD.
- 32 eFisioTrack: a telerehabilitation environment based on motion recognition using
- 33 accelerometry. ScientificWorldJournal. 2014;12: 495391. doi:
- 34 10.1155/2014/495391.
- 35 20. García J, Ruiz D, Soriano A, Marin O, Hernandez-Sanchez S, Ferrairaó S.
- 36 eFisioTrack: A Telerehabilitation Platform for Monitoring Prescribed
- 37 Therapeutic Exercises in Orthopaedic Injuries. In: Ambient Assisted Living and
- Home Care. Lecture Notes in Computer Science. Volume 7657, 2012, pp 423-430.
- 39 21. Beaton DE, Davis AM, Hudak P, McConnell S. The DASH (Disabilities of the Arm,
- Shoulder and Hand) outcome measure: What do we know about it now? Br J Hand
- 41 Ther. 2001; 6(4): 109-118. doi.org/10.1177/175899830100600401

- 22. Hervás MT, Navarro A, Peidró S, Rodrigo JL, López P, Martínez I. Spanish version of the DASH questionnaire. Cross-cultural adaptation, reliability, validity and responsiveness. Med Clin (Barc) 2006; 127(12): 441-447.
- 23. Tate AR, McClure PW, Young IA, Salvatori R, Michener LA. Comprehensive impairment based exercise and manual therapy intervention for patients with subacromial impingement syndrome: a case series. The Journal of Orthoaedic and Sports Physical Therapy 2010; 40(8): 474-493. doi: 10.2519/jospt.2010.3223.
- 24. Franchignoni F, Vercelli S, Giordano A, Sartorio F, Bravini E, Ferriero G. Minimal clinically important difference of the disabilities of the arm, shoulder and hand outcome measure (DASH) and its shortened version (QuickDASH). J Orthop Sports Phys Ther 2014; 44(1): 30-39. doi: 10.2519/jospt.2014.4893
- 25. Roy JS, MacDermid JC, Woodhouse LJ. A systematic review of the psychometric properties of the Constant-Murley score. J Shoulder Elbow Surg 2010;19(1):157-164. doi: 10.1016/j.jse.2009.04.008.
- 26. Bankes MJ, Emery RJ. An evaluation of the Constant-Murley shoulder assessment.
   J Bone Joint Surg Br. 1997;79(4):696.
- 27. Kitis A, Celik E, Aslan UB, Zencir M. DASH questionnaire for the analysis of musculoskeletal symptoms in industry workers: a validity and reliability study.

  Journal of Applied Ergonomics 2009; 40(2): 251-255. doi: 10.1016/j.apergo.2008.04.005.
- 28. Pastora- Bernal JM, Martín-Valero R, Barón-López FJ, Moyan N, Estebanez-Pérez MJ. Telerehabilitation after arthroscopic subacromial decompression is effective and not inferior to standard practice: Preliminary results. J Telemed Telecare. 2018a;24(6):428-433. doi: 10.1177/1357633X17706583.
- 29. Dias Correia F, Molinos M, Luis S, Carvalho D, Carvalho C, Costa P, Seabra R,
   Francisco G, Bento V, Lains J. Digitally assisted conventional home-based rehabilitation after arthroscopic rotarot cuff repair: a randomized controlled trial. Am
   J Phys Med Rehabil. 2022;101(3):237-249. doi:10.1097/PHM.0000000000001780.
- 30. Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res 1987; 214: 160-164.
- 31. Grassi FA, Tajana MS. The normalization of data in the Constant-Murley score for 32 the shoulder. A study conducted on 563 healthy subjects. Chir Organi Mov. 2003; 33 88(1):65-73.
- 32. Kachingwe AF, Philips B, Sletten E, Plunkett SW. Comparison of manual therapy techniques with therapeutic exercise in the treatment of shoulder impingement: a randomized controlled pilot clinical trial. J Man Manip Ther 2008;16(4):238-47.doi: 10.1179/106698108790818314.
- 33. Lombardi I, Magri AG, Fleury AM, Da Silva AC, Natour J. Progressive resistance training in patients with shoulder impingement syndrome: a randomized controlled trial. Arthritis Rheum. 2008;59(5):615-22. doi: 10.1002/art.23576.

- 1 34. Seron P, Oliveros MJ, Gutierrz-Areias R, Fuentes-Aspe R, Torres-Castro RC,
- 2 Merino-Osorio C, Nahuelhual P, Inostroza J, Jalil Y, Solano R, Marzuca-Nassr GN,
- 3 Agulera-Eguia R, Lavados-Romo P, Soto-Rodríguez FJ, Sabelle C, Villarroel-Silve
- 4 G, Gomolan P, Huaiquilaf S, Sanchez P. Effectiveness of Telerehabilitation in
- 5 Physical Therapy: A Rapid Overview. Phys Ther 2021;101(6):pzab053. doi:
- 6 10.1093/ptj/pzab053.
- 7 35. Muñoz-Tomás MT, Burillo-Lafuente M, Vicente-Parra A, Sanz-Rubio MC, Suarez-
- 8 Serrano C, Marcén-Román Y, Franco-Sierra MA. Telerehabilitation as a Therapeutic
- 9 Exercise Tool versus Face-to-Face Physiotherapy: A Systematic Review. Int J
- 10 Environ Res Public Health. 2023;20(5):4358. doi: 10.3390/ijerph20054358.
- 36. Muscillo R. Schmid M, Conforto S, D'Alessio T. Early recognition of upper limb
- motor tasks through accelerometers: real-time implementation of a DTW-based
- 13 algorithm. Comput Biol Med 2011; 41(3): 164-172. doi:
- 14 10.1016/j.compbiomed.2011.01.007.
- 15 37. Huang K, Sparto PJ, Kiesler S, Siewiorek DP, Smailagic A. iPod-based in-home
- system for monitoring gaze-stabilization exercise compliance of individuals with
- vestibular hypofunction. J NeuroEng Rehab 2014, 11:69. doi: 10.1186/1743-0003-
- 18 11-69.
- 19 38. Tao G, Miller WC, Eng JJ, Esfandiari E, Imam B, Lindstrom H, Payne MW. Group-
- 20 based telerehabilitation intervention using Wii Fit to improve walking in older adults
- with lower limb amputation (WiiNWalk): A randomized control trial. Clin Rehabil.
- 22 2022;36(3):331-341. doi: 10.1177/02692155211061222.
- 23 39. Yuen HK, Lowman JD, Oster RA, de Andrade JA. Home-Based Pulmonary
- Rehabilitation for Patients With Idiopathic Pulmonary Fibrosis: a pilot study. J
- 25 Cardiopulm Rehabil Prev. 2019;39(4):281-284. doi:
- 26 10.1097/HCR.0000000000000418.
- 40. Essery R, Geraghthy A, Kirby S, Yardley. Predictors of adherence to home-based
- physical therapies: a systematic review. Disabil Rehabil. 2017;39(6):519-534.doi:
- 29 10.3109/09638288.2016.1153160.
- 30 41. Himler P, Lee GT, Rhon DI, Young JL, Cook C, Rentmeester C. Understanding
- barriers to adherence to home exercise programs in patients with musculoskeletal
- neck pain. Musculoskelet Sci Pract. 2023;63:102722. doi:
- 33 10.1016/j.msksp.2023.102722.
- 34 42. Palazzo C, Klinger E, Dorner V, Kadri A, Thierry O, Boumenir Y, Martin W,
- Poiraudeau S, Ville I. Barriers to home-based exercise program adherence with
- 36 chronic low back pain: Patient expectations regarding new technologies. Ann Phys
- 37 Rehabil Med. 2016;59(2):107-13.doi: 10.1016/j.rehab.2016.01.009.
- 43. Jirasakulsuk N, Saengpromma P, Khruakhorn. Real-Time Telerehabilitation in Older
- 39 Adults With Musculoskeletal Conditions: Systematic Review and Meta-analysis.
- 40 JMIR Rehabil Assist Technol 2022;9(3):e36028.doi: 10.2196/36028.
- 41 44. Belotti N, Bonfantil S, Locatelli A, Rota L, Ghidotti A, Vitali A. A Tele-
- 42 Rehabilitation Platform for Shoulder Motor Function Recovery Using Serious

- Games and an Azure Kinect Device. Stud Health Technol Inform. 2022 May 16;293:145-152. doi: 10.3233/SHTI220361.
- 45. Gava V, Ribeiro LP, Barreto R, Rezende C. Effectiveness of physical therapy given by telerehabilitation on pain and disability of individuals with shoulder pain: A
  - systematic review. Clin Rehabil. 2022;36(6):715-725. doi:
- 6 10.1177/02692155221083496.
- 46. Eriksson L, Lindström B, Gard G, et al. Physiotherapy at a distance: a controlled study of rehabilitation at home after a shoulder joint operation. J Telemed Telecare 2009; 15(5): 215–220. doi: 10.1258/jtt.2009.081003.
- 47. Jordan JL, Holden MA, Mason EE, Foster NE. Interventions to improve adherence to exercise for chronic musculoskeletal pain in adults. Cochrane Database Syst Rev 2010(1); 20: CD005956. doi:10.1002/14651858.CD005956.
- 48. Pastora-Bernal JM, Martín-Valero R, Barón-López FJ. Cost analysis of
   telerehabilitation after arthroscopic subacromial decompression. J Telemed Telecare.
   2018b;24(8):553-559. doi: 10.1177/1357633X17723367.
- 49. Kloek C, van Dongen J, de Baker D, Bossen D, Dekker J, Veenhof C. Cost-effectiveness of a blended physiotherapy intervention compared to usual physiotherapy in patients with hip and/or knee osteoarthritis: a cluster randomized controlled trial. BMC Public Health. 2018;18(1):1082.doi: 10.1186/s12889-018-
- 20 5975-7.

- 50. Nelson M, Russell T, Crossley K, Bourke M, McPhail. Cost-effectiveness of telerehabilitation versus traditional care after total hip replacement: A trial-based economic evaluation. J Telemed Telecare. 2019;27(6):359-366.doi: 10.1177/1357633X19869796.
- 51. Fatoye F, Gebrye T, Fatoye C, Mbada ChE, Olaoye MI, Odolr AC, Dada O. The
   Clinical and Cost-Effectiveness of Telerehabilitation for People With Nonspecific
   Chronic Low Back Pain: Randomized Controlled Trial. JMIR Mhealth
- 28 Uhealth. 2020;8(6):e15375. doi: 10.2196/15375.
- 52. Torpil B, Kaya Ö. The Effectiveness of Client-Centered Intervention With
   Telerehabilitation Method After Total Knee Arthroplasty. OTJR (Thorofare N
   J). 2022;42(1):40-49. doi: 10.1177/15394492211038293.
- 53. Suso-Martí L, La Touche R, Herranz-Gómez A, Díaz-Parreño SA, París-Alemnay
   A, Cuenca-Martínez F. Effectiveness of Telerehabilitation in Physical Therapist
   Practice: An Umbrella and Mapping Review With Meta-Meta-Analysis. Phys
   Ther. 2021;101(5):pzab075. doi: 10.1093/ptj/pzab075.
- 54. Dueñas L, Aguilar-Rodríguez M, Voogt L, Lluch E, Struyf F, Mertens M, De
   Meulemeester K, Meeus M. Specific versus Non-Specific Exercises for Chronic
   Neck or Shoulder Pain: A Systematic Review. J Clin Med. 2021;10(24):5946.doi:
- 39 10.3390/jcm10245946.











# INFORMED CONSENT FOR PARTICIPATION IN THE PROJECT OF MONITORING SHOULDER REHABILITATION EXERCISES WITH THE EFISIOTRACK SYSTEM

| Mr./Mrs | | |
|---|---|---|
| | . as a patient, being years old, resid | ng at |
| I DECLARE THAT: | | |
| The physiotherapi | ist | , has explained |

#### 1.- Identification, description and objectives of the procedure.

Bioinspired Health Engineering group of the University of Alicante, in collaboration with the Physiotherapy area of the Miguel Hernández University of Elche and the General University Hospital of Elche, intends to carry out a study on exercise monitoring for shoulder rehabilitation with inertial sensors located in a game console (Wii) controller. This controller is connected to a computer and allows you to record the exercises you perform, as well as their trajectory and speed. The physiotherapist who treats you, will be able to see in real time from another location, if you complete the prescriptions that have been made, as well as interact with you if necessary through videoconference.

The results obtained will serve to refine the system and generalize its application to the population that performs therapeutic exercise for shoulder injuries and needs follow-up on them.

The procedure that is proposed to me consists of placing a movement sensor attached to the extremities or the trunk (depending on the exercise) with a velcro so that it registers how the exercise is performed. Everything will be visible on a screen, which will provide information on the range of movement of the exercise, the repetitions and series that you have to do, as well as if you are executing them correctly.

#### 2.- Benefits that are expected to be achieved

I will not receive any financial compensation or other benefits for being evaluated. In any case, if the research were successful, it could help to perfect the system and extend its use as an aid to carrying out home exercise programs (without specialist supervision).

#### 3.- Reasonable alternatives

The decision to participate in the work or to complete the data on the evaluation *is completely voluntary*, and I may refuse to receive it and may even revoke my consent at any time, without having to give any explanation and without prejudice to my personal consideration.











#### 4.- Foreseeable consequences of its performance and non-performance

If I <u>freely and voluntarily</u> decide to carry out the eccentric work protocol and be evaluated later, I will have the right to decide whether or not to be informed of the results of the investigation, if it is finally carried out.

#### 5.- Frequent and infrequent risks

No harmful risks are expected since the system will record movement during therapeutic exercise and does not modify its characteristics or parameters at all.

# 6.- Risks and consequences depending on the personal clinical situation of the patient and their personal or professional circumstances . None

# 7.- Protection of personal data and confidentiality.

The information about my personal and health data will be incorporated and processed in a computerized database, complying with the guarantees established la Leyfor the Protection of Personal Data and health legislation.

The assignment to other research centers will be carried out through a disassociation procedure through which an identification code will be generated that prevents me from being directly or indirectly identified.

Likewise, I have been informed that I have the possibility of exercising the *rights of access*, *rectification, cancellation and opposition to the processing of personal data*, in the terms provided in the applicable regulations.

If you decide to revoke the consent that I now give, the data obtained from the examination at that time will continue to be part of the research.

# 8.- Project manager

The person in charge of the research project is Dr. Antonio Soriano Payá, professor in the Department of Information Technology and Computing at the University of Alicante











# Therefore, having read the above information, <u>I understand that</u>:

My participation in this study is voluntary, and I can revoke my consent at any time, without explanation and without affecting my medical care.

I give my consent for la Universidad MiguelHernández or other research centers to use my data, including my health information, for medical research, always maintaining my anonymity and the confidentiality of my data.

The information and this document have been provided to me sufficiently in advance to reflect calmly and make my decision freely and responsibly.

I have understood the explanations that have been provided to me in clear and simple language and the physiotherapist who has treated me has allowed me to make all the observations and has clarified all the doubts that I have raised.

confidentiality of these data will be maintained in accordance with the provisions of Organic Law 15/1999 on the Protection of Personal Data. In addition, the confidentiality of clinical data will be maintained according to LAW 41/2002, of November 14, the basic regulation of patient autonomy and rights and obligations regarding clinical information and documentation.

Observations you consider making:











Therefore, I state that I am satisfied with the information received and under such conditions I agree and CONSENT to participate in the study on 'Monitoring for the performance of therapeutic rehabilitation exercises'

| (Name and two surnames) (Name and two surnames) (Name and two surnames) | | |
|---|---|---|
| Signed.: | Signed | Signed: |
| Signature of the patient Signature of a witness Signature of the Physiotherapist | | |
| In Date | e: (day)/ (month)/ (year) | |

RESPONSIBLE FOR THE PROJECT

Dr. Antonio Soriano Payá











# **REVOCATION OF INFORMED CONSENT**

| Mr./Mrs. as a patient |
|---|
| (or representative of the patient D), of |
| ID. nº I revoke the consent given on date, which I end with this date and without having to give explanations. |
| In of of 20 |
| Signature of the patient Signature of a witness Signature of the Physiotherapist ID: |
| Signed: Signed: Signed: |
| (Name and two surnames) (Name and two surnames) (Name and two surnames) |